CLINICAL TRIAL: NCT00481065
Title: A Phase II, Randomized, Controlled, Open Label, Single-Center Study to Evaluate the Immunogenicity, Safety and Tolerability of an H5N1-vaccine and a Seasonal Influenza Vaccine in Adult Subjects
Brief Title: Immunogenicity, Safety and Tolerability of Prepandemic Influenza and Seasonal Influenza Vaccine in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V87P5
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Pandemic; Avian Influenza
Keywords: Bird flu; influenza vaccine; Seasonal influenza vaccine; Prepandemic vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

ARMS (8):
- Concomitant alone (Experimental): 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1 then 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382.
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- Concomitant +Mixed (Experimental): 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1, 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- Concomitant +MF59-eH5N1 (Experimental): 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1, 1 dose of MF59-eH5N1 on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- Mixed (Experimental): 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 1 and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- Mixed and mixed (Experimental): 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 1, day 22, and day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- Mixed+MF59-eH5N1 (Experimental): 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 1, 1 dose of MF59-eH5N1 on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- MF59-eH5N1+eTIV_a (Experimental): 1 dose of MF59-eH5N1 on day 1, 1 dose of eTIV_a on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a
- eTIV_a+MF59-eH5N1 (Experimental): 1 dose of eTIV_a on day 1, 1 dose of MF59-eH5N1 on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
  Interventions: Biological: MF59-eH5N1; Biological: eTIV_a; Biological: MF59-eH5N1 + eTIV_a

INTERVENTIONS:
Biological: MF59-eH5N1
Biological: eTIV_a
Biological: MF59-eH5N1 + eTIV_a

SUMMARY:
This study evaluates the immunogenicity, safety and tolerability of an H5N1 vaccine with a seasonal trivalent influenza vaccine, containing the strains recommended by WHO for the 2007 influenza season in the Southern Hemisphere.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 405 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Drug Information Services +1 800 244 7668, Study Chair — Novartis
Locations (1):
- Bogotá, Colombia

REFERENCES:
- [Result] Lopez P, Caicedo Y, Sierra A, Tilman S, Banzhoff A, Clemens R. Combined, concurrent, and sequential administration of seasonal influenza and MF59-adjuvanted A/H5N1 vaccines: a phase II randomized, controlled trial of immunogenicity and safety in healthy adults. J Infect Dis. 2011 Jun 15;203(12):1719-28. doi: 10.1093/infdis/jir191. PMID 21606530
- [Derived] Lopez P, Caicedo Y, Sierra A, Tilman S, Clemens R, Banzhoff A. Combined administration of MF59-adjuvanted A/H5N1 prepandemic and seasonal influenza vaccines: long-term antibody persistence and robust booster responses 1 year after a one-dose priming schedule. Clin Vaccine Immunol. 2013 May;20(5):753-8. doi: 10.1128/CVI.00626-12. Epub 2013 Mar 27. PMID 23536690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 center in Colombia.
Pre-assignment Details: All subjects enrolled were included in the trial. A total of 405 subjects was enrolled and randomized into 8 groups in this study. The participant flow data are from the all randomized set.
Groups:
- Concomitant Alone: 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1 then 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1 then 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
- Concomitant+Mixed: 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1, 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
- Concomitant+MF59-eH5N1: 1 dose of MF59-eH5N1 into one arm and 1 dose of eTIV_a into the other arm on day 1, 1 dose of MF59-eH5N1 on day 22, and 1 dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 382
- Mixed + Mixed: dose of MF59-eH5N1 mixed extemporaneously with eTIV_a on day 1, day 22, and day 382
Period: Overall Study
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Started | 51 | 50 | 51 | 52 | 51 | 51 | 50 | 49
Completed | 29 | 33 | 32 | 37 | 28 | 27 | 34 | 30
Not Completed | 22 | 17 | 19 | 15 | 23 | 24 | 16 | 19
Not completed — Adverse event or death | 1 | 1 | 3 | 0 | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 11 | 12 | 7 | 11 | 13 | 12 | 9 | 10
Not completed — Lost to Follow-up | 4 | 2 | 4 | 3 | 3 | 3 | 2 | 5
Not completed — Inappropriate enrollment | 4 | 0 | 2 | 0 | 2 | 1 | 0 | 1
Not completed — Administrative reason | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 1 | 1 | 2 | 6 | 3 | 2
Not completed — Unable to classify | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The demographic characteristics of the randomized population are summarized in this section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1 | Total
Number analyzed (Participants) | 51 | 50 | 51 | 52 | 51 | 51 | 50 | 49 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6.2) | 29.4 (5.8) | 29.5 (6.5) | 29.8 (6.8) | 29.6 (6.1) | 28.8 (6.2) | 27.9 (6.2) | 30.1 (6.2) | 29.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 31 | 36 | 30 | 36 | 39 | 30 | 32 | 276
  Male | 9 | 19 | 15 | 22 | 15 | 12 | 20 | 17 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number Subjects Who Responded to Two or Three Vaccinations of the MF59-H5N1 Influenza Vaccine
Description: Seroconversion (serocon.) is defined as negative pre-vaccination serum (titer <10 for HI [Haemagglutination Inhibition], area ≤4 mm^2 for SRH [Single Radial Haemolysis]) / positive post-vaccination titer (titer ≥ 40 for HI, area ≥ 25 mm^2 for SRH).
  Significant increase in antibody titer is defined as at least a fourfold increase from non-negative pre-vaccination serum (HI ≥ 10) or at least 50% increase in the SRH area.
  Seroprotection is defined as a HI titer ≥40 and a SRH area ≥25 mm^2.
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Population: The analysis was done on the full analysis set (FAS).
Measure: Number; unit: Subjects
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Subjects
  HI seroprot. (day1) N=46,48,47,50,49,48,48,44 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
  HI serocon. (2nd vacc) N=46,48,46,49,48,48,47,43 | 12 [14 to 41] | 33 [54 to 81] | 37 [66 to 91] | 13 [15 to 41] | 31 [49 to 78] | 34 [56 to 83] | 19 [26 to 56] | 22 [35 to 67]
  HI seroprot. (2nd vacc) N=46,48,46,49,48,48,47,43 | 12 [14 to 41] | 34 [56 to 83] | 37 [66 to 91] | 14 [17 to 43] | 32 [52 to 80] | 34 [56 to 83] | 19 [26 to 56] | 22 [35 to 67]
  HI serocon. (3rd vacc) N=23,24,36,39,31,20,32,32 | 17 [52 to 90] | 15 [39 to 79] | 26 [76 to 99] | 19 [37 to 71] | 16 [43 to 82] | 13 [41 to 85] | 24 [67 to 96] | 16 [43 to 82]
  HI seroprot. (3rd vacc) N=24,25,28,35,25,20,28,25 | 18 [53 to 90] | 15 [39 to 79] | 26 [76 to 99] | 20 [39 to 74] | 16 [43 to 82] | 14 [46 to 88] | 24 [67 to 96] | 16 [43 to 82]
  SRH seroprot. (day 1) N=46,48,47,50,49,48,48,44) | 3 | 6 | 1 | 4 | 4 | 6 | 4 | 5
  SRH serocon. (2nd vacc) N=46,48,46,50,46,48,47,42 | 14 [18 to 46] | 38 [65 to 90] | 43 [82 to 99] | 11 [12 to 37] | 31 [52 to 80] | 38 [67 to 91] | 23 [34 to 64] | 25 [43 to 74]
  SRH seroprot. (2nd vacc) N=46,48,46,50,48,48,47,43 | 17 [23 to 52] | 40 [70 to 93] | 43 [82 to 99] | 14 [16 to 42] | 35 [58 to 85] | 42 [75 to 95] | 26 [40 to 70] | 29 [51 to 81]
  SRH serocon. (3rd vacc) N=25,25,28,35,25,20,28,25 | 24 [80 to 100] | 20 [59 to 93] | 27 [82 to 100] | 27 [54 to 85] | 12 [28 to 69] | 12 [36 to 81] | 18 [44 to 81] | 16 [43 to 82]
  SRH seroprot. (3rd vacc) N=25,25,28,35,25,20,28,25 | 25 [86 to 100] | 21 [64 to 95] | 27 [82 to 100] | 27 [60 to 90] | 11 [24 to 65] | 15 [51 to 91] | 23 [63 to 94] | 19 [55 to 91]
  MN ≥40 (day 1) N=46,48,47,50,49,48,48,44) | 11 | 11 | 10 | 11 | 10 | 10 | 11 | 11
  MN ≥40 (2nd vacc) N=46,48,46,50,48,48,47,43 | 14 [18 to 46] | 36 [60 to 86] | 44 [85 to 99] | 16 [20 to 47] | 36 [60 to 86] | 44 [80 to 98] | 24 [36 to 66] | 20 [31 to 62]
  MN ≥40 (3rd vacc) N=25,25,28,35,25,20,28,25 | 24 [80 to 100] | 24 [80 to 100] | 28 [88 to 100] | 31 [73 to 97] | 22 [69 to 97] | 20 [83 to 100] | 26 [76 to 99] | 23 [74 to 99]

2. Primary Outcome: Geometric Mean Ratio After Two or Three Vaccinations of the MF59-eH5N1 Influenza Vaccine
Description: Geometric mean Ratio (GMR) was calculated for the haemagglutination inhibition (HI), microneutralization (MN) and single-radial haemolysis (SRH) result as well as the associated 95% confidence intervals. GMR was calculated as 21 days after second and third vaccinations over day 1.
Time Frame: 21 days after second and third vaccinations (day 22 and day 43)
Population: Full analysis set (FAS)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Ratio
  HI (2nd vacc) N= 46,48,46,49,48,48,47,43 | 2.11 [1.29 to 3.46] | 12 [7.09 to 19] | 23 [14 to 37] | 2.16 [1.33 to 3.49] | 9.52 [5.86 to 15] | 14 [8.32 to 22] | 2.96 [1.81 to 4.86] | 5.34 [3.2 to 8.91]
  HI (3rd vacc) N= 24,25,28,35,25,20,28,25 | 34 [15 to 76] | 17 [7.82 to 37] | 93 [44 to 197] | 10 [5.36 to 20] | 9.89 [4.5 to 22] | 21 [8.56 to 49] | 66 [31 to 139] | 12 [5.53 to 26]
  SRH (2nd vacc) N= 46,48,46,49,46,47,47,42 | 1.82 [1.35 to 2.44] | 5.32 [3.98 to 7.09] | 9.64 [7.17 to 13] | 1.58 [1.19 to 2.11] | 4.25 [3.16 to 5.71] | 6.04 [4.5 to 8.11] | 2.9 [2.16 to 3.88] | 3.26 [2.39 to 4.44]
  SRH (3rd vacc) N= 25,25,28,35,25,20,28,25 | 9.92 [6.73 to 15] | 6.22 [4.25 to 9.12] | 11 [7.47 to 16] | 5.13 [3.69 to 7.13] | 3.1 [2.07 to 4.65] | 6.76 [4.33 to 11] | 7.17 [4.95 to 10] | 4.55 [3.08 to 6.74]
  MN (2nd vacc) N= 46,48,47,50,49,48,48,44 | 2.12 [1.54 to 2.91] | 7.64 [5.61 to 10] | 13 [9.45 to 18] | 2.15 [1.59 to 2.92] | 6.79 [4.98 to 9.26] | 11 [8.04 to 15] | 3.86 [2.82 to 5.29] | 3.49 [2.52 to 4.84]
  MN (3rd vacc) N= 24,25,28,35,25,20,28,25 | 38 [23 to 64] | 39 [23 to 64] | 66 [40 to 109] | 16 [10 to 25] | 13 [8 to 23] | 23 [13 to 41] | 58 [36 to 95] | 21 [12 to 35]

3. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions by Vaccination
Description: The evaluate the safety of the administration of two or three vaccinations of MF59-eH5N1 influenza vaccine, either given sequentially, concomitantly or mixed extemporaneously with seasonal eTIV_a influenza vaccine.
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Measure: Number; unit: Subjects
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 50 | 50 | 51 | 51 | 51 | 50 | 49 | 49
Subjects
  Erythema (N=50,48,47,51,48,47,47,43) 2nd vacc | 0 | 8 | 8 | 0 | 8 | 8 | 7 | 5
  Induration (N=50,48,47,51,48,47,47,43) 2nd vacc | 0 | 2 | 3 | 0 | 3 | 2 | 1 | 3
  Swelling (N=50,48,47,51,48,47,47,43) 2nd vacc | 0 | 2 | 5 | 0 | 4 | 1 | 1 | 1
  Ecchymosis (N=50,48,47,51,48,47,47,43) 2nd vacc | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Pain (N=50,48,47,51,48,47,47,43) 2nd vacc | 0 | 21 | 16 | 0 | 20 | 18 | 12 | 16
  Erythema (N=31,33,36,39,31,29,34,31) 3rd vacc | 8 | 4 | 9 | 9 | 0 | 7 | 6 | 11
  Induration (N=31,33,36,39,31,29,34,31) 3rd vacc | 6 | 6 | 14 | 9 | 0 | 9 | 7 | 8
  Swelling (N=31,33,36,39,31,29,34,31) 3rd vacc | 5 | 3 | 9 | 2 | 0 | 8 | 6 | 5
  Ecchymosis (N=31,33,36,39,31,29,34,31) 3rd vacc | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 3
  Pain (N=31,33,36,39,31,29,34,31) 3rd vacc | 20 | 16 | 21 | 23 | 20 | 0 | 17 | 15
  Chills (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 0 | 1 | NA — Vaccine was not administered on this date. | 2 | 4 | 2 | 2
  Malaise (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 2 | 4 | NA — Vaccine was not administered on this date. | 7 | 6 | 2 | 6
  Myalgia (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 8 | 7 | NA — Vaccine was not administered on this date. | 9 | 6 | 3 | 5
  Arthralgia (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 0 | 3 | NA — Vaccine was not administered on this date. | 1 | 4 | 2 | 2
  Headache (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 2 | 5 | NA — Vaccine was not administered on this date. | 6 | 5 | 3 | 4
  Sweating (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 0 | 1 | NA — Vaccine was not administered on this date. | 0 | 2 | 1 | 1
  Fatigue (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 1 | 0 | NA — Vaccine was not administered on this date. | 1 | 1 | 2 | 2
  Nausea (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 0 | 1 | NA — Vaccine was not administered on this date. | 1 | 1 | 2 | 2
  Fever≥ 38°C (N=50,48,47,51,48,47,47,43) 2nd vacc | NA — Vaccine was not administered on this date. | 0 | 0 | NA — Vaccine was not administered on this date. | 1 | 3 | 0 | 2
  Chills (N=31,49,36,39,31,50,34,49) 3rd vacc | 3 | 0 | 6 | 3 | 4 | 0 | 3 | 0
  Malaise (N=31,33,36,39,31,29,34,32) 3rd vacc | 6 | 5 | 9 | 10 | 8 | 7 | 9 | 7
  Myalgia (N=30,33,36,39,31,29,34,32) 3rd vacc | 12 | 11 | 17 | 13 | 12 | 10 | 8 | 13
  Arthralgia (N=31,33,36,39,31,29,34,32) 3rd vacc | 2 | 0 | 5 | 4 | 4 | 3 | 4 | 4
  Headache (N=31,32,36,39,31,29,34,32) 3rd vacc | 8 | 7 | 11 | 7 | 10 | 8 | 5 | 7
  Sweating (N=31,49,36,39,51,29,49,32) 3rd vacc | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 3
  Fatigue (N=31,33,36,39,31,50,34,32) 3rd vacc | 2 | 1 | 3 | 1 | 2 | 2 | 1 | 1
  Nausea (N=31,33,36,39,31,50,34,32) 3rd vacc | 1 | 1 | 3 | 2 | 3 | 0 | 2 | 2
  Fever≥ 38°C (N=31,48,47,51,48,29,34,32) 3rd vacc | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2

4. Primary Outcome: Number of Subjects Who Responded to Two Vaccinations of the Seasonal eTIV_a Influenza Vaccines (Strain H1N1)
Description: seroconversion: negative pre-vaccination serum (HI titer <10, SRH area =<4 mm^2)/positive post-vaccination titer (HI titer =>10) or at least 50% increase in the SRH area.
  Seroprotection is defined as a HI titer ≥40 and a SRH area ≥25 mm^2.
Time Frame: 21 days after second vaccination (day 43)
Population: The analysis was done on the full analysis set (FAS).
Measure: Number; unit: Subjects
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Subjects
  HI seroprot. (day 1) | 13 | 18 | 16 | 23 | 15 | 19 | 24 | 20
  HI seroconversion N=46,48,46,49,48,48,47,43 | 33 [57 to 84] | 35 [58 to 85] | 36 [64 to 89] | 29 [43 to 72] | 37 [63 to 88] | 37 [63 to 88] | 29 [46 to 75] | 31 [56 to 85]
  HI seroprotection N=46,48,46,49,48,48,47,43 | 37 [66 to 91] | 45 [83 to 99] | 43 [82 to 99] | 39 [64 to 88] | 44 [80 to 98] | 41 [72 to 94] | 43 [80 to 98] | 40 [81 to 99]

5. Primary Outcome: Number of Subjects Who Responded to Two or Three Vaccinations of the Seasonal eTIV_a Influenza Vaccines (Strain H3N2)
Description: seroconversion (serocon.): negative pre-vaccination serum (HI titer <10, SRH area =<4 mm^2)/positive post-vaccination titer (HI titer =>10) or at least 50% increase in the SRH area.
  Seroprotection is defined as a HI titer ≥40 and a SRH area ≥25 mm^2.
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Population: The analysis was done on the full analysis set (FAS).
Measure: Number; unit: Subjects
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Subjects
  HI seroprot. (day 1) | 20 | 22 | 14 | 23 | 26 | 22 | 12 | 22
  HI serocon. (2nd vacc) N=46,48,46,49,48,48,47,43 | 23 [35 to 65] | 36 [60 to 86] | 35 [61 to 87] | 35 [55 to 82] | 40 [70 to 93] | 40 [70 to 93] | 35 [60 to 86] | 29 [51 to 81]
  HI seroprot. (2nd vacc) N=46,48,46,50,48,48,47,43) | 39 [71 to 94] | 46 [86 to 99] | 44 [85 to 99] | 49 [89 to 100] | 48 [93 to 100] | 48 [93 to 100] | 47 [92 to 100] | 40 [81 to 99]
  HI serocon. (3rd vacc) N=25,25,28,35,25,20,28,25 | 19 [55 to 91] | 20 [59 to 93] | 26 [76 to 99] | 30 [70 to 95] | 18 [51 to 88] | 17 [62 to 97] | 25 [72 to 98] | 21 [64 to 95]
  HI seroprot. (3rd vacc) N=30,33,36,39,31,29,34,32 | 18 [53 to 90] | 15 [39 to 79] | 26 [76 to 99] | 20 [39 to 74] | 16 [43 to 82] | 14 [46 to 88] | 86 [67 to 96] | 64 [43 to 82]

6. Primary Outcome: Number of Subjects Who Responded to Two or Three Vaccinations of the Seasonal eTIV_a Influenza Vaccines (Strain B)
Description: as for outcome 5
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Population: The analysis was done on the full analysis set (FAS).
Measure: Number; unit: Subjects
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Subjects
  HI seroprot. (day 1) | 5 | 4 | 6 | 10 | 2 | 9 | 12 | 5
  HI serocon. (2nd vacc) N=46,48,46,50,48,48,47,43 | 37 [66 to 91] | 38 [65 to 90] | 36 [64 to 89] | 41 [69 to 91] | 41 [72 to 94] | 35 [58 to 85] | 36 [62 to 88] | 28 [49 to 79]
  HI seroprot. (2nd vacc) N=46,48,46,50,48,48,47,43 | 40 [74 to 95] | 43 [77 to 97] | 42 [79 to 98] | 46 [81 to 98] | 44 [80 to 98] | 45 [83 to 99] | 44 [82 to 99] | 32 [59 to 86]
  HI serocon. (3rd vacc) N=25,25,28,35,25,20,28,25 | 19 [55 to 91] | 17 [46 to 85] | 19 [48 to 84] | 27 [60 to 90] | 15 [39 to 79] | 13 [41 to 85] | 11 [22 to 59] | 15 [39 to 79]
  HI seroprot. (3rd vacc) N=25,25,28,35,25,20,28,25 | 22 [69 to 97] | 21 [64 to 95] | 22 [59 to 92] | 31 [73 to 97] | 18 [51 to 88] | 18 [68 to 99] | 17 [41 to 78] | 20 [59 to 93]

7. Primary Outcome: Geometric Mean Ratio After Two Doses of the Seasonal eTIV_a Influenza Vaccine (Strain H1N1)
Description: For each vaccine group, the least squares GMRs were calculated for the haemagglutination inhibition (HI) results as well as the associated 95% confidence intervals. GMR was calculated over day 1.
Time Frame: 21 days after second vaccination (day 43)
Population: Full analysis set (FAS)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 46 | 50 | 48 | 48 | 47 | 43
Ratio | 15 [9.54 to 23] | 13 [8.43 to 20] | 14 [8.82 to 21] | 6.77 [4.46 to 10] | 12 [7.81 to 18] | 10 [6.69 to 16] | 6.23 [4.03 to 9.61] | 11 [6.76 to 17]

8. Secondary Outcome: Number of Subjects With Immunogenicity Results After the Booster Vaccination Against the MF59-eH5N1 Influenza Vaccine Mixed Extemporaneously With the Seasonal eTIV_a Influenza Vaccine
Description: Booster was given on day 382; seroconversion: negative pre-vaccination serum (HI titer <10, SRH area ≤ 4 mm^2)/positive post-vaccination titer (HI titer ≥10) or at least 50% increase in SRH area; Seroprotection is defined as a HI titer ≥40 and a SRH area ≥25 mm^2.
  The number of subjects achieving seroconversion or significant increase and seroprotection were calculated at day 382.
Time Frame: 21 days after booster vaccination (day 403)
Population: Full analysis set (FAS)
Measure: Number; unit: Subjects
Arm/Group | Mixed | Mixed + Mixed
Number analyzed (Participants) | 39 | 31
Subjects
  Seroprotection (HI) _MF59-H5N1 (N=35, 25) | 26 [57 to 88] | 16 [43 to 82]
  Seroconversion (HI)_MF59-H5N1 | 25 [54 to 85] | 15 [39 to 79]
  Seroprotection (SRH)_MF59-H5N1 (N=35, 25) | 50 [39 to 74] | 7 [12 to 49]
  Seroconversion (SRH)_MF59-H5N1 (N=35, 25) | 21 [42 to 76] | 10 [21 to 61]
  Seroprotection (HI) - eTIV_a (H1N1) N=35, 25 | 33 [81 to 99] | 24 [80 to 100]
  Seroconversion (HI) - eTIV_a (H1N1) N=39, 25 | 17 [31 to 66] | 10 [21 to 61]
  Seroprotection (HI) - eTIV_a (H3N2) N=35, 25 | 35 [90 to 100] | 25 [86 to 100]
  Seroconversion (HI) - eTIV_a (H3N2) N=39, 25 | 12 [19 to 52] | 5 [7 to 41]
  Seroprotection (HI) - eTIV_a (B) N=35, 25 | 31 [73 to 97] | 18 [51 to 88]
  Seroconversion (HI) - seTIV_a (B) N=35, 25 | 6 [7 to 34] | 4 [5 to 36]

9. Primary Outcome: Geometric Mean Ratio After Two or Three Vaccinations of the Seasonal eTIV_a Influenza Vaccine (Strain H3N1)
Description: For each vaccine group, the least squares GMRs were calculated for the haemagglutination inhibition (HI) results for each time point of the study, as well as the associated 95% confidence intervals. GMR was calculated over day 1.
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Population: Full analysis set (FAS)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Ratio
  HI GMR (2nd vacc) N= 46,48,46,50,48,48,47,43 | 6.01 [4.01 to 9.01] | 9.72 [6.54 to 14] | 9.34 [6.22 to 14] | 11 [7.54 to 16] | 11 [7.26 to 16] | 10 [6.92 to 15] | 11 [7.25 to 16] | 7.54 [4.96 to 11]
  HI GMR (3rd vacc) N= 25,25,28,35,25,20,28,25 | 17 [9.56 to 29] | 10 [6.04 to 18] | 17 [9.86 to 28] | 18 [11 to 29] | 8.92 [5.12 to 16] | 11 [5.8 to 20] | 17 [10 to 29] | 13 [7.64 to 23]

10. Primary Outcome: Geometric Mean Ratio After Two or Three Vaccinations of the Seasonal eTIV_a Influenza Vaccine (Strain B)
Description: as for outcome 9
Time Frame: 21 days after second and third vaccinations (day 43 and day 403)
Population: Full analysis set (FAS)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Number analyzed (Participants) | 46 | 48 | 47 | 50 | 49 | 48 | 48 | 44
Ratio
  HI GMR (2nd vacc) N= 46,48,46,50,48,48,47,43 | 11 [7.85 to 17] | 13 [9.01 to 19] | 10 [6.94 to 15] | 10 [7.22 to 15] | 17 [12 to 25] | 8.77 [6.07 to 13] | 10 [6.97 to 15] | 8.0 [5.44 to 12]
  HI GMR (3rd vacc) N= 25,25,28,35,25,20,28,25 | 8.85 [5.86 to 13] | 5.47 [3.64 to 8.22] | 7.95 [5.37 to 12] | 7.17 [5.05 to 10] | 5.29 [3.51 to 8] | 5.1 [3.22 to 8.06] | 4.17 [2.82 to 6.18] | 4.26 [2.84 to 6.4]

11. Secondary Outcome: Geometric Mean Ratio After the Booster Vaccination Against the MF59-eH5N1 Influenza Vaccine Mixed Extemporaneously With the Seasonal eTIV_a Influenza Vaccine
Description: For each vaccine group, the least squares GMRs were calculated for the HI and SRH results for each time point of the study, as well as the associated 95% confidence intervals. GMR was calculated over day 382 for all time points for the booster dose.
Time Frame: 21 days after booster vaccination (day 403)
Population: Full analysis set (FAS)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mixed | Mixed + Mixed
Number analyzed (Participants) | 39 | 31
Ratio
  HI (MF59-H5N1) N=35, 25 | 13 [6.99 to 25] | 7.14 [3.4 to 15]
  SRH (MF59-H5N1) N=35, 25 | 4.88 [3.59 to 6.63] | 2.77 [1.93 to 3.98]
  HI (eTIV_a, H1N1) N=35, 25 | 4.82 [3.05 to 7.73] | 2.61 [1.51 to 4.51]
  HI (eTIV_a, H3N2) N=35, 25 | 2.62 [1.83 to 3.76] | 2.21 [1.44 to 3.39]
  HI (eTIV_a, B) N=35, 25 | 1.96 [1.55 to 2.48] | 1.94 [1.47 to 2.55]

ADVERSE EVENTS:
Time Frame: All adverse events and serious adverse events were collected for 20 months (the duration of the study).
Description: the number of subjects included here are from the safety population and not the enrolled population as disclosed in the Demography and Study Termination sections.
Arm/Group | Concomitant Alone | Concomitant+Mixed | Concomitant+MF59-eH5N1 | Mixed | Mixed + Mixed | Mixed+MF59-eH5N1 | MF59-eH5N1+eTIV_a | eTIV_a+MF59-eH5N1
Serious Adverse Events (participants affected / at risk) | 4/50 | 1/50 | 2/51 | 3/51 | 3/51 | 0/50 | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 38/50 | 42/50 | 41/51 | 39/51 | 42/51 | 43/50 | 37/49 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Alone (N=50) | Concomitant+Mixed (N=50) | Concomitant+MF59-eH5N1 (N=51) | Mixed (N=51) | Mixed + Mixed (N=51) | Mixed+MF59-eH5N1 (N=50) | MF59-eH5N1+eTIV_a (N=49) | eTIV_a+MF59-eH5N1 (N=49)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration bronchial (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
B-Cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Alone (N=50) | Concomitant+Mixed (N=50) | Concomitant+MF59-eH5N1 (N=51) | Mixed (N=51) | Mixed + Mixed (N=51) | Mixed+MF59-eH5N1 (N=50) | MF59-eH5N1+eTIV_a (N=49) | eTIV_a+MF59-eH5N1 (N=49)
Gastritis (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 2 | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 5 | 6 | 2 | 5 | 4 | 4 | 7
Chills (General disorders) | 5 | 5 | 10 | 8 | 8 | 8 | 5 | 3
Fatigue (General disorders) | 3 | 4 | 5 | 3 | 5 | 4 | 4 | 4
Injection site erythema (General disorders) | 12 | 17 | 17 | 16 | 21 | 16 | 16 | 21
Injection site haemorrhage (General disorders) | 3 | 5 | 2 | 5 | 5 | 3 | 3 | 3
Injection site induration (General disorders) | 11 | 15 | 20 | 16 | 15 | 15 | 10 | 15
Injection site pain (General disorders) | 29 | 34 | 33 | 32 | 34 | 32 | 33 | 29
Injection site swelling (General disorders) | 8 | 9 | 13 | 10 | 10 | 10 | 9 | 11
Malaise (General disorders) | 15 | 17 | 21 | 19 | 20 | 21 | 17 | 13
Pyrexia (General disorders) | 5 | 0 | 1 | 4 | 4 | 8 | 2 | 6
Influenza (Infections and infestations) | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Tonsillitis (Infections and infestations) | 2 | 2 | 0 | 0 | 2 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 9 | 6 | 6 | 9 | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 24 | 24 | 23 | 22 | 17 | 18 | 17
Headache (Nervous system disorders) | 18 | 15 | 22 | 14 | 25 | 19 | 13 | 15
Migraine (Nervous system disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 4 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 8 | 4 | 3 | 4 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days